CLINICAL TRIAL: NCT04095377
Title: Development of Automated Analysis to Electroencephelogram (EEG) Data in Patients Treated at the Sagol Hyperbaric Medicine and Research Center at the Years 2017-2019 - A Retrospective Study
Brief Title: Development of Automated Analysis to Electroencephelogram (EEG) Data in Patients Treated at the Sagol Hyperbaric Medicine and Research Center at the Years 2017-2019.
Status: Completed | Type: Observational
Sponsor: QuantalX Neuroscience (Industry)
Responsible Party: Sponsor
Other Study IDs: 0292-18
Record Dates: First submitted 2019-03-25; First posted 2019-09-19 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2019-03

CONDITIONS: Healthy; CVA; Hemorrhage; TBI (Traumatic Brain Injury); Concussion, Brain; Fibromyalgia; ABD; Adhd; Dementia; Mci; Cognitive Impairment; Cognitive Decline; MS (Multiple Sclerosis)
MeSH Terms: conditions — Hemorrhage; Brain Injuries, Traumatic; Brain Concussion; Fibromyalgia; Attention Deficit Disorder with Hyperactivity; Dementia; Neurocognitive Disorders; Cognitive Dysfunction; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (13):
- healthy
  Interventions: Other: No intervention, this is a retrospective study.
- CVA
  Interventions: Other: No intervention, this is a retrospective study.
- Hammorhage
  Interventions: Other: No intervention, this is a retrospective study.
- TBI
  Interventions: Other: No intervention, this is a retrospective study.
- Concussion
  Interventions: Other: No intervention, this is a retrospective study.
- Fibromyalgia
  Interventions: Other: No intervention, this is a retrospective study.
- ABD
  Interventions: Other: No intervention, this is a retrospective study.
- ADHD
  Interventions: Other: No intervention, this is a retrospective study.
- MCI
  Interventions: Other: No intervention, this is a retrospective study.
- DEMENTIA
  Interventions: Other: No intervention, this is a retrospective study.
- COGNITIVE IMPAIRMENT
  Interventions: Other: No intervention, this is a retrospective study.
- COGNITIVE DECLINE
  Interventions: Other: No intervention, this is a retrospective study.
- MS
  Interventions: Other: No intervention, this is a retrospective study.

INTERVENTIONS:
Other: No intervention, this is a retrospective study. — No intervention, this is a retrospective study.

SUMMARY:
DELPhI software developed for the analysis of EEG recordings in response to magnetic stimulation in relation to clinical data.

DETAILED DESCRIPTION:
Collection of EEG data, recorded at Sagol center for hyperbaric medicine and research in the years of 2017-2019 of patients arriving to be treated at the hyperbaric chamber before,during and after treatments. EEG was recorded of patients during cognitive tests, resting state and during magnetic stimulation as a part of other array of tests performed at the Sagol center. Anonymous EEG data along with MRI scans, PET-CT, SPECT, cognitive tests, Medical history and medications will be transferred to QuantalX Neuroscience LTD.

QuantalX Neuroscience is intending to use the above mentioned data in order to improve DELPhI, an algorithm for the analysis of EEG recordings in response to magnetic stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over the age of 18.
* Subjects that performed at least one EEG test as a part of their hyperbaric treatment at Sagol center Asaf-Harophe.

Exclusion Criteria:

* Subjects with no EEG test or that their EEG recording is in pure quality, not allowing analysis of the data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient arriving to be treated at the Sagol center for hyperbaric medicine and research at Asaf-Harophe in te years of 2017-2019.
Sampling Method: Non-Probability Sample
Enrollment: 875 (Actual)
Dates: Start 2019-03-24 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Defining Plasticity (the ratio between excitatory to inhibitory brain response) Means and STD in each cohort. | through study completion, an average of 1 year
  Measure of the mean and STD Plasticity of each cohort.
Defining Connectivity (dispersion of brain signal) Means and STD in each cohort. | through study completion, an average of 1 year
  Measure of the mean and STD Connectivity of each cohort.
Defining Plasticity (the ratio between excitatory to inhibitory brain response) standard error (SEM) in each cohort. | through study completion, an average of 1 year
  Measure of the standard error (SEM) of Plasticity of each cohort.
Defining Connectivity (dispersion of brain signal) standard error (SEM) in each cohort. | through study completion, an average of 1 year
  Measure of the standard error (SEM) of Connectivity of each cohort.
Defining Plasticity (excitation/inhibition brain response) coefficient of variation (CV%) in each cohort. | through study completion, an average of 1 year
  Measure of the coefficient of variation (CV%) of Plasticity of each cohort.
Defining Connectivity (dispersion of brain signal) coefficient of variation (CV%) in each cohort. | through study completion, an average of 1 year
  Measure of the coefficient of variation (CV%) of Connectivity of each cohort.
Defining Plasticity (excitation/inhibition brain response) minimum, median, maximum in each cohort. | through study completion, an average of 1 year
  Measure of the minimum, median, maximum of Plasticity of each cohort.
Defining Connectivity (dispersion of brain signal) minimum, median, maximum in each cohort. | through study completion, an average of 1 year
  Measure of the minimum, median, maximum of Connectivity of each cohort.
Defining Plasticity (excitation/inhibition brain response) 95% confidence interval in each cohort. | through study completion, an average of 1 year
  Measure of the 95% confidence interval of Plasticity of each cohort.
Defining Connectivity (dispersion of brain signal) 95% confidence interval in each cohort. | through study completion, an average of 1 year
  Measure of the 95% confidence interval of Connectivity of each cohort.

CONTACTS AND LOCATIONS:
Locations (1):
- Asaf-Harophe, Rishon LeZiyyon, Israel

IPD SHARING:
Plan to Share IPD: Undecided